CLINICAL TRIAL: NCT04046380
Title: A Modified Mathematical Model to Calculate Power Received by Mechanically Ventilated Patients With Different Etiologies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Deng Kuo, Doctor, Changhua Christian Hospital
Other Study IDs: 108-CCH-IRP-081
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Acute Respiratory Distress Syndrome, Mechanical Ventilation, Respiratory Mechanics, Ventilator-induced Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal lungs
  Interventions: Diagnostic Test: work of breath measurement and calculation
- Acute respiratory distress syndrome (ARDS) group
  Interventions: Diagnostic Test: work of breath measurement and calculation

INTERVENTIONS:
Diagnostic Test: work of breath measurement and calculation — The ventilator-imposed power at various tidal volume (6, 8, 10 ml/Kg) and positive end-expiratory pressure (5, 10 cmH 2 O) will be calculated by the formula.

SUMMARY:
Ventilator-induced lung injury is a common complication. The latest and most noticeable theory of its pathogenesis is called 'ergotrauma' by Gattinoni in 2016. The theory uses ventilator-imposed 'energy' or 'power' to encompass several known forms of injury-inducing factors such as pressure,volume, flow, rate, etc. However, to quantify power imposed by ventilator is no easy task in clinical practice. So, Gattinoni proposed a mathematical formula for easy power calculation. However, Gattinoni did not compare the difference between various etiologies of acute lung injury. We will enroll 100 patients (50 with acute respiratory distress syndrome and 50 with normal lung). The ventilator-imposed power at various tidal volume (6, 8, 10 ml/Kg) and positive end-expiratory pressure (5, 10 cmH2O) will be calculated by the formula. The area enclosed by hysteresis of pressure-volume curve, and hence the work it implies, will be measured as a standard. Our study will aim to compare the formula in different patient groups and in Taiwanese people.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients aged 20 to 90 years old

Exclusion Criteria:

* Fraction of inspired oxygen (FiO2) higher than 60%
* Acute physiology and chronic health evaluation (APACHE) II score more than 30
* Plateau pressure or peak airway pressure more than 30 cmH2O
* High risk for barotrauma
* Unstable hemodynamic status
* Under airway pressure release ventilation or high frequency oscillation ventilation therapy
* Under extra-corporeal membrane oxygenation support
* On prone position

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single ICU in one teaching hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
correlation of calculated and measured work of breath | The measurement and calculation will be performed only once when the ventilator was in use. The estimated time frame of measurement is less than one hour.
  The ventilator-imposed power at various tidal volume (6, 8, 10 ml/Kg) and positive end-expiratory pressure (5, 10 cmH 2 O) will be calculated by the formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Oba Y, Salzman GA. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury. N Engl J Med. 2000 Sep 14;343(11):813; author reply 813-4. No abstract available. PMID 10991706
- [Background] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Background] Gattinoni L, Marini JJ, Collino F, Maiolo G, Rapetti F, Tonetti T, Vasques F, Quintel M. The future of mechanical ventilation: lessons from the present and the past. Crit Care. 2017 Jul 12;21(1):183. doi: 10.1186/s13054-017-1750-x. PMID 28701178
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Tonetti T, Vasques F, Rapetti F, Maiolo G, Collino F, Romitti F, Camporota L, Cressoni M, Cadringher P, Quintel M, Gattinoni L. Driving pressure and mechanical power: new targets for VILI prevention. Ann Transl Med. 2017 Jul;5(14):286. doi: 10.21037/atm.2017.07.08. PMID 28828361